CLINICAL TRIAL: NCT05470322
Title: Efficacy and Tolerability of a Fractional Ablative Erbium Laser for Axillary Scarring for Hidradenitis Suppurativa Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients were able to consented/enrolled into the study during the period of time the study was approved by the IRB. Study officially withdrawn with the IRB on 11/24/2025.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-14262
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Hidradenitis Suppurativa; Scarring
MeSH Terms: conditions — Hidradenitis Suppurativa; Cicatrix | interventions — Lasers, Solid-State; Lasers

STUDY DESIGN:
Masking Description: No masking will be performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Laser Treatment (Experimental): The parameters of the laser will be set according to optimal operation protocol and in accordance with guidelines set forth by Sciton. Each laser treatment will take approximately 10 to 15 minutes per subject to target HS scarring.
  Interventions: Device: Er: YAG laser

INTERVENTIONS:
Device: Er: YAG laser — Patients will be treated with laser for their HS scarring.
  Other Names: laser; fractional ablative laser

SUMMARY:
Single center, open-label, baseline-controlled study evaluating the use of a Sciton fractionated ablative laser in the treatment of Hidradenitis Suppurativa (HS) scarring.

DETAILED DESCRIPTION:
Single center, open-label, baseline-controlled study evaluating the use of a Sciton fractionated ablative laser in the treatment of Hidradenitis Suppurativa (HS) scarring. The device is FDA approved for the treatment of scarring in all skin types. The study team seeks to observe the efficacy and tolerability in patients without active HS lesions. The study may enroll up to 19 subjects looking for improvement in their HS scarring in the axillary region. The subjects will receive treatment with the Sciton Joule Er:YAG 2940nm laser along with treatment with topical tretinoin, hydroquinone, and hydrocortisone starting 1 month prior to first laser treatment as per standard of care for scar treatment. Each patient will receive 3 treatments spaced approximately one month apart. The patients will be surveyed about their quality of life due to HS scarring, as well as their perspectives on their axillary scarring before and after their assigned treatments. All patients included in the study will have no contraindications to either laser or the use of standard treatment protocol (tretinoin and hydroquinone). Subjects in the laser group will complete a DLQI (Dermatology Life Quality Index) survey, patient satisfaction survey, and clinical photographs at each treatment visit and at follow-up 1, 2, and 3 months after the last treatment. Subjects in the topical treatment group will be evaluated at the initial visit, month 3 and month 6.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females, ≥ 18 years of age at time of informed consent with no upper age limit, seeking treatment for HS scarring in the axillary region.
* Subjects must voluntarily sign and date an IRB approved informed consent form.
* Subjects with diagnosis of HS (Hidradenitis Suppurativa) scarring recorded over the past 6 months.
* Subject has an HS PGA (Hidradenitis Suppurativa Physician's Global Assessment) Scale of 0 or 1
* Able to read, understand and voluntarily provide written informed consent.
* Subjects are determined to be healthy, non-smokers.
* Subjects able and willing to comply with the treatment protocol and follow-up schedule and requirements.
* Understand and accept the obligation not to undergo any other procedures in the areas to be treated through the follow-up period.

Exclusion Criteria:

* Subject does not have the capacity to consent to the study.
* Subject underwent any medical-grade scar treatments (ie, lasers, excision procedures, topical prescriptions for scars) in the past 6 months prior to enrollment in the study.
* Any history of keloid scarring.
* Any previous surgical procedure in the treatment area in the past 12 months, or major surgery in the last 6 months.
* History of immunosuppression/immune deficiency disorders (including AIDS and HIV infection), and/or any history of systemic chemotherapy for prior 12 months.
* Subject has no health contraindications to receiving local lidocaine and epinephrine injections, including but not limited to any form of heart disease or arrhythmia, untreated or uncontrolled severe hypertension, uncontrolled hyperthyroidism, uncontrolled diabetes, pheochromocytoma, Cocaine use.
* History or current use of the following prescription medications:Accutane or other systemic retinoids within the past twelve months, Tricyclic antidepressant, monoamine oxidase inhibitors, B-blocker
* Smoking or vaping in the past 12 months.
* History of an allergy or an adverse reaction to hydroquinone or tretinoin.
* History of photosensitivity and/or connective tissue disease.
* History of uncontrolled diabetes, hypertension and depression.
* History of ongoing pregnancy, active breastfeeding, cancer, and epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Modified Scale for HS Scar Severity (mSHSS) | Month 0
  HS Scar Severity will be assessed in participants using mSHSS as follows:
  Clear - 0 - No visible scars from HS Almost Clear -1 - Hardly visible from 2.5 m away Mild - 2-Easily recognizable; less than half the affected area Moderate - 3 - More than half the affected area involved Severe - 4 - Entire area involved Very Severe - 5 - Entire area with prominent atrophic or hypertrophic scars
Modified Scale for HS Scar Severity (mSHSS) | Month 6
  HS Scar Severity will be assessed in participants using mSHSS as follows:
  Clear - 0 - No visible scars from HS Almost Clear -1 - Hardly visible from 2.5 m away Mild - 2-Easily recognizable; less than half the affected area Moderate - 3 - More than half the affected area involved Severe - 4 - Entire area involved Very Severe - 5 - Entire area with prominent atrophic or hypertrophic scars

SECONDARY OUTCOMES:
Subject Satisfaction Survey | Month 1
  Following treatment participants will be asked to complete a survey in the clinic while referring to their image in a mirror and comparing post-treatment photos versus baseline photos. Scoring will be assessed as follows (-3 = Greatly decreased, -2 = Moderately decreased, -1 = Slightly decreased, 0 = No change, 1 = Slightly increased, 2 = Moderately increased, 3 = Greatly increased) with a lower overall score denoting improvement in appearance.
Subject Satisfaction Survey | Month 2
  Following treatment participants will be asked to complete a survey in the clinic while referring to their image in a mirror and comparing post-treatment photos versus baseline photos. Scoring will be assessed as follows (-3 = Greatly decreased, -2 = Moderately decreased, -1 = Slightly decreased, 0 = No change, 1 = Slightly increased, 2 = Moderately increased, 3 = Greatly increased) with a lower overall score denoting improvement in appearance.
Subject Satisfaction Survey | Month 3
  Following treatment participants will be asked to complete a survey in the clinic while referring to their image in a mirror and comparing post-treatment photos versus baseline photos. Scoring will be assessed as follows (-3 = Greatly decreased, -2 = Moderately decreased, -1 = Slightly decreased, 0 = No change, 1 = Slightly increased, 2 = Moderately increased, 3 = Greatly increased) with a lower overall score denoting improvement in appearance.
Subject Satisfaction Survey | Month 4
  Participants will be asked to complete a survey in the clinic while referring to their image in a mirror and comparing post-treatment photos versus baseline photos. Scoring will be assessed as follows (-3 = Greatly decreased, -2 = Moderately decreased, -1 = Slightly decreased, 0 = No change, 1 = Slightly increased, 2 = Moderately increased, 3 = Greatly increased) with a lower overall score denoting improvement in appearance.
Subject Satisfaction Survey | Month 5
  Participants will be asked to complete a survey in the clinic while referring to their image in a mirror and comparing post-treatment photos versus baseline photos. Scoring will be assessed as follows (-3 = Greatly decreased, -2 = Moderately decreased, -1 = Slightly decreased, 0 = No change, 1 = Slightly increased, 2 = Moderately increased, 3 = Greatly increased) with a lower overall score denoting improvement in appearance.
Subject Satisfaction Survey | Month 6
  Participants will be asked to complete a survey in the clinic while referring to their image in a mirror and comparing post-treatment photos versus baseline photos. Scoring will be assessed as follows (-3 = Greatly decreased, -2 = Moderately decreased, -1 = Slightly decreased, 0 = No change, 1 = Slightly increased, 2 = Moderately increased, 3 = Greatly increased) with a lower overall score denoting improvement in appearance.
Physician graded assessment of scar severity | Month 0
  Scar severity will be assessed in participants by way of GAIS (Global Aesthetic Improvement Scale) using photographic assessments. Scoring will range from -3 (greatly worsened scar severity) to 3 (greatly improved scar severity). A score of zero represents no change in scar severity.
Physician graded assessment of hyperpigmentation | Month 0
  Hyperpigmentation will be assessed in participants by way of GAIS (Global Aesthetic Improvement Scale) using photographic assessments. Scoring will range from -3 (greatly worsened hyperpigmentation) to 3 (greatly improved hyperpigmentation). A score of zero represents no change in hyperpigmentation.
Physician graded assessment of scar severity | Month 2
  Scar severity will be assessed in participants by way of GAIS (Global Aesthetic Improvement Scale) using photographic assessments. Scoring will range from -3 (greatly worsened scar severity) to 3 (greatly improved scar severity). A score of zero represents no change in scar severity.
Physician graded assessment of hyperpigmentation | Month 2
  Hyperpigmentation will be assessed in participants by way of GAIS (Global Aesthetic Improvement Scale) using photographic assessments. Scoring will range from -3 (greatly worsened hyperpigmentation) to 3 (greatly improved hyperpigmentation). A score of zero represents no change in hyperpigmentation.
Physician graded assessment of scar severity | Month 3
  Scar severity will be assessed in participants by way of GAIS (Global Aesthetic Improvement Scale) using photographic assessments. Scoring will range from -3 (greatly worsened scar severity) to 3 (greatly improved scar severity). A score of zero represents no change in scar severity.
Physician graded assessment of hyperpigmentation | Month 3
  Hyperpigmentation will be assessed in participants by way of GAIS (Global Aesthetic Improvement Scale) using photographic assessments. Scoring will range from -3 (greatly worsened hyperpigmentation) to 3 (greatly improved hyperpigmentation). A score of zero represents no change in hyperpigmentation.
Physician graded assessment of scar severity | Month 4
  Scar severity will be assessed in participants by way of GAIS (Global Aesthetic Improvement Scale) using photographic assessments. Scoring will range from -3 (greatly worsened scar severity) to 3 (greatly improved scar severity). A score of zero represents no change in scar severity.
Physician graded assessment of hyperpigmentation | Month 4
  Hyperpigmentation will be assessed in participants by way of GAIS (Global Aesthetic Improvement Scale) using photographic assessments. Scoring will range from -3 (greatly worsened hyperpigmentation) to 3 (greatly improved hyperpigmentation). A score of zero represents no change in hyperpigmentation.
Physician graded assessment of scar severity | Month 5
  Scar severity will be assessed in participants by way of GAIS (Global Aesthetic Improvement Scale) using photographic assessments. Scoring will range from -3 (greatly worsened scar severity) to 3 (greatly improved scar severity). A score of zero represents no change in scar severity.
Physician graded assessment of hyperpigmentation | Month 5
  Hyperpigmentation will be assessed in participants by way of GAIS (Global Aesthetic Improvement Scale) using photographic assessments. Scoring will range from -3 (greatly worsened hyperpigmentation) to 3 (greatly improved hyperpigmentation). A score of zero represents no change in hyperpigmentation.
Physician graded assessment of hyperpigmentation | Month 6
  Hyperpigmentation will be assessed in participants by way of GAIS (Global Aesthetic Improvement Scale) using photographic assessments. Scoring will range from -3 (greatly worsened hyperpigmentation) to 3 (greatly improved hyperpigmentation). A score of zero represents no change in hyperpigmentation.
Physician graded assessment of scar severity | Month 6
  Scar severity will be assessed in participants by way of GAIS (Global Aesthetic Improvement Scale) using photographic assessments. Scoring will range from -3 (greatly worsened scar severity) to 3 (greatly improved scar severity). A score of zero represents no change in scar severity.

CONTACTS AND LOCATIONS:
Overall Officials: Kseniya Kobets, MD, Principal Investigator — Albert Einstein College of Medicine Montefiore Medical Center
Locations (1):
- Montefiore Einstein Advanced Care, Elmsford, New York, United States

IPD SHARING:
Plan to Share IPD: No